CLINICAL TRIAL: NCT06163222
Title: Can User-centred Design and Behavioural-science Informed Interventions Improve Equity in Outpatient Access in North West London? A Non-randomised Controlled Trial
Brief Title: Behavioural Interventions to Improve Equity in Outpatient Access
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23IC8361
Record Dates: First submitted 2023-11-21; First posted 2023-12-08 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Behavioural Science Interventions to Improve Health Equity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Getting to your appointment (Experimental): Additional 14-day message reminder that includes link to new transport index web page
  Interventions: Behavioral: Additional message with behavioural science-informed content and associated web pages
- Help with travel costs (Experimental): Additional 14-day message reminder that includes link to new 'help with travel costs' web page
  Interventions: Behavioral: Additional message with behavioural science-informed content and associated web pages
- What to expect (Experimental): Additional 14-day message reminder that includes link to 'what to expect' web page
  Interventions: Behavioral: Additional message with behavioural science-informed content and associated web pages
- Usual communications (Active Comparator): Existing communication strategy used for each of the five clinical specialties e.g. reminder messages 3 and 7 days prior to outpatient appointment
  Interventions: Other: Usual communication strategy

INTERVENTIONS:
Behavioral: Additional message with behavioural science-informed content and associated web pages — Behavioural science-informed messages sent 14-days prior to outpatient appointment which include links to re-designed web pages
  Arms: Getting to your appointment; Help with travel costs; What to expect
Other: Usual communication strategy — Usual communications sent from outpatient services to remind participants about their appointments
  Arms: Usual communications

SUMMARY:
The goal of this clinical trial is to improve health equity within outpatient service access. This is through design and behavioural science-informed interventions that aim to improve rates of first outpatient appointment attendance. Health equity refers to the avoidable and unfair differences in health access, outcomes and experience between groups or populations. Outpatient services are those appointments where advice from a specialised medical professional is provided to a patient in a clinic setting.

This clinical trial aims to test different ways of supporting people to attend their first outpatient appointments at five clinical specialties (ophthalmology, gastroenterology, colorectal surgery, cardiology and plastic surgery) at Imperial College Healthcare NHS Trust (ICHT). It is specifically focused on improving attendance for people who are most likely to miss their appointment based on ICHT data, which includes people from minority ethnic backgrounds and people living in the most deprived postcodes.

The main question this clinical trial aims to answer is:

• Do behavioural science-informed message interventions improve rates of first outpatient appointment attendance in patients facing inequity of access based on ethnicity and deprivation?

The secondary questions this clinical trial aims to answer include:

* Do behavioural science-informed message interventions improve rates of first outpatient appointment attendance across all patient groups?
* Do behavioural science-informed message interventions increase the number of patients who "self-cancel" their appointment if they need to?
* In which patient groups did the message interventions have most impact, e.g., a certain age range?
* Which factors were associated with improved outpatient attendance rates specifically in participants from minority ethnic groups or living in area with highest level of deprivation?
* What was the overall outcome of all first outpatient appointments included in the clinical trial?
* What was the overall successful message delivery rate for the messages sent as part of the study? Were there particular participant groups that were more likely to have an undelivered message?
* What was the overall outcome of appointment attendance for people who received a text message intervention compared with receiving a text message and/or email intervention?
* How well did participants engage with the message interventions e.g. did they click the link provided in the message?

DETAILED DESCRIPTION:
This clinical trial has been designed as a non-randomised controlled trial, aiming to test the impact of three design and behavioural science-informed interventions on first outpatient appointment attendance in groups at highest risk of inequity. The interventions will be tested in five clinical specialties at ICHT - cardiology, gastroenterology, ophthalmology, plastic surgery, and colorectal surgery. The study is estimated to last 48 weeks. The messages sent as part of the trial will be deployed by ICHT staff members who manage outpatient services.

Prior to conducting this trial, three message and web page interventions were co-designed with a diverse group of public members with good representation from the IMD and ethnicity groups facing inequity of access, ICHT staff, researchers, and behavioural science experts. These interventions were based on insights on barriers to appointment attendance gained from short qualitative interviews conducted with people who had missed appointments at ICHT and who also faced inequity based on ethnicity or deprivation.

This study has been designed to have four arms. These four arms will include a control arm, that will be the standard practice communication strategy used by each clinical specialty, as well as three intervention strategies. Currently the standard communications that patients receive before an outpatient appointment varies, but commonly patients receive a reminder 3 and 7 days before the appointment at ICHT. The three co-designed interventions for the trial are all based on an additional message reminder to this existing reminder schedule that will be sent to patients 14 days before their appointment. DrDoctor is the message provider that is currently used by ICHT and that the interventions will be housed in. The web pages will be housed in the existing ICHT website. All five clinical specialties will spend one week in each study arm, before cycling to the next arm. They will move from one arm to the next, until they return to their original study arm, resulting in continuous four-week cycles until the final study period is reached. Therefore, the five clinical specialties will all be in the same study arms at the same time and go through the cycle together until the sample size is reached. This method of allocation of clinics to study arms has been selected as it is not possible with the current technology being used at ICHT to randomise participants within clinics to different study arms.

Data will be collected on the message delivery and appointment outcomes throughout the trial and full analysis will take place at the end of the trial, once the sample size has been reached. The rate of missed appointments will be monitored throughout the study to assess if there is any backfire effect of the interventions.

For the first approximately 20 weeks of the study, only participants who received the intervention as a text message will be analysed. However after this point, as email notifications were turned on by ICHT for all patients, both text and/or email interventions will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have been referred to their first outpatient appointment at one of five ICHT adult clinical specialties - Cardiology, Colorectal Surgery, Gastroenterology, Ophthalmology and Plastic Surgery.

Exclusion Criteria:

* Phone or video appointments
* Diagnostics appointments
* Two-week wait appointments
* Saturday or Sunday appointments
* Appointments without message reminders switched on in DrDoctor
* Patients who re-enter the study and receive >1 intervention
* Patients who received email message reminders about their appointment (until 23rd May 2024, after which they will be included due to change in ICHT communications approach)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13389 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Change in Did Not Attend (DNA) rate for first outpatient appointment across five clinical specialties with an emphasis on participants' ethnicity and the deprivation level of their address (Index of Multiple Deprivation quintiles) | End of study period (12 months)
  Did Not Attend (DNA) rate is the change over time in the number of people who do not attend their outpatient appointment without cancelling or rescheduling. This rate will be analysed for the clinics included in the study and to see if it changes over time with our interventions.
  While this change in DNA rate over time will be analysed for all patients, the research team will focus particularly on how this changes with a patient's ethnicity and the deprivation of where they live. Deprivation is currently recorded by ICHT using the Index of Multiple Deprivation (IMD) which assigns a score to a patient's postcode to indicate its level of deprivation based on multiple factors.

SECONDARY OUTCOMES:
Change in DNA rate at first outpatient appointment across all five clinical specialties for all participant groups | End of study period (12 months)
  Did Not Attend (DNA) rate is the change over time in the number of people who do not attend their outpatient appointment without cancelling or rescheduling. This rate will be analysed for the clinics included in the study and to see if it changes over time with our interventions.
  While the primary outcome focuses on ethnicity and deprivation, this outcome will focus on describing any other changes in DNA rate seen across all patient groups.
Change in Patient-Initiated Cancellation (PIC) rate for first outpatient appointment across all five clinical specialties. | End of study period (12 months)
  Patient-Initiated Cancellation (PIC) rate is the change over time in the number of people who cancel their outpatient appointment ahead of time. This rate will be analysed for the clinics included in the study and to see if it changes over time with our interventions.
Change in DNA rate at first outpatient appointment across all five clinical specialties for population subgroups, controlling for variables such as ethnicity, participant demographics, clinic specialty and IMD | End of study period (12 months)
  Did Not Attend (DNA) rate is the change over time in the number of people who do not attend their outpatient appointment without cancelling or rescheduling.
  This will provide an evaluation of where the selected interventions had most impact according to patient characteristics. Focus will be given to analysing in more detail patients of 'Black', 'mixed' or 'other' ethnicity as well as those living in areas with the greatest level of deprivation (IMD quintile 1) to further understand what variables are associated with a decrease in DNA rates in these populations specifically.
Change in the rate of appointment outcomes (attended, DNA, PIC, Hospital-Initiated Cancellation) for first outpatient appointments across all five clinical specialties | End of study period (12 months)
  Analysis will be carried out to understand what the outcomes of all appointments included in the study and how this changes from the start of the study. For example, the outcomes could be that the patient attended the appointment, missed the appointment, cancelled the appointment in advance or the hospital cancelled the appointment.
Differences between message delivery rate for study interventions across all five clinical specialties for different population subgroups | End of study period (12 months)
  The study team will analyse the message delivery rate for the study interventions. This refers to the number of messages that were successfully delivered to study participants. This will be analysed to see if unsuccessful message delivery rates are associated with specific population subgroups e.g. patients living in more deprived areas.
Differences between each study intervention's click-through rate from message to web page for all participant groups | End of study period (12 months)
  The click-through rate for the study interventions will be analysed as part of the study, which describes the proportion of people who click the link provided in the messages as part of the study to view the associated web page. The different interventions will be compared to see which had higher click-through rates over time.
Differences between each study intervention's web page engagement using Google Analytics for each of the study interventions for all participant groups | End of study period (12 months)
  The Google Analytics report for the ICHT web pages developed as part of the study will be analysed to understand which parts of the pages that people engaged with most and how they interacted with the site, a tool and practice that is currently already used at ICHT. The different web pages reports will be compared with each other to review their engagement over time.
Change in the rate of appointment outcomes (attended, DNA, PIC, Hospital-Initiated Cancellation) for appointments that received text message-only and appointments that received text and/or email interventions | End of study period (12 months)
  For the first approximately 20 weeks of the study, data will be analysed for appointments that received text message-only interventions. This is because only a small number of patients had opted into email reminders, so these patients were going to be removed for analysis. However, ICHT turned on automatic email notifications for all patients during the study, and after this stage both text message and email reminders will be analysed. The study team will analyse appointment attendance between people who received just the text message interventions compared with people who received text and email interventions, once ICHT had turned on email reminders.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Huf, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers.

REFERENCES:
- [Background] Huf S, Kerrison RS, King D, Chadborn T, Richmond A, Cunningham D, Friedman E, Shukla H, Tseng FM, Judah G, Darzi A, Vlaev I. Behavioral economics informed message content in text message reminders to improve cervical screening participation: Two pragmatic randomized controlled trials. Prev Med. 2020 Oct;139:106170. doi: 10.1016/j.ypmed.2020.106170. Epub 2020 Jun 29. PMID 32610059
- [Background] Acharya A, Ashrafian H, Cunningham D, Ruwende J, Darzi A, Judah G. Evaluating the impact of a novel behavioural science informed animation upon breast cancer screening uptake: protocol for a randomised controlled trial. BMC Public Health. 2022 Jul 19;22(1):1388. doi: 10.1186/s12889-022-13781-x. PMID 35854267
- [Background] Hallsworth M, Berry D, Sanders M, Sallis A, King D, Vlaev I, Darzi A. Stating Appointment Costs in SMS Reminders Reduces Missed Hospital Appointments: Findings from Two Randomised Controlled Trials. PLoS One. 2015 Sep 14;10(9):e0137306. doi: 10.1371/journal.pone.0137306. eCollection 2015. PMID 26366885
- See also: NHS England. Core20PLUS5 (adults) - an approach to reducing healthcare inequalities [Internet]. 2023 [cited 2023 Nov 17]. — http://www.england.nhs.uk/about/equality/equality-hub/national-healthcare-inequalities-improvement-programme/core20plus5/#:~:text=Core20PLUS5%20is%20a%20national%20NHS,clinical%20areas%20requiring%20accelerated%20improvement